CLINICAL TRIAL: NCT05750095
Title: Enabling Parents of Children With Autism Spectrum Disorders - a Randomized Controlled Trial of Parenting Programs
Acronym: ENACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Helse Fonna (Other); St. Olavs Hospital (Other); University of Bergen (Other); Norwegian University of Science and Technology (Other); NORCE Norwegian Research Centre AS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2899
Record Dates: First submitted 2023-01-26; First posted 2023-03-01 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-01

CONDITIONS: Autism Spectrum Disorder
Keywords: Stress; Parenting; Autism
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — First Aid

STUDY DESIGN:
Masking Description: All measures are parent reported
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Incredible Years Autism Spectrum and Language Delay Programme (Experimental): Incredible Years Autism Spectrum and Language Delay Programme is a manualised group based intervention in 13 weekly 2-hour sessions. The programme targets parents of children aged 2-6 years, with autism spectrum disorder or language delay.
  Interventions: Behavioral: Incredible Years Autism Spectrum and Language Delay Programme
- First Aid for Parents (Active Comparator): "First Aid for Parents" is a program consisting of three full day work-shops targeting communication, interaction and daily living skills for parents of children with autism spectrum disorders
  Interventions: Behavioral: First Aid for Parents

INTERVENTIONS:
Behavioral: Incredible Years Autism Spectrum and Language Delay Programme — Incredible Years Autism Spectrum and Language Delay Programme is a manualised group based intervention in 13 weekly 2-hour sessions. The programme targets parents of children aged 2-6 years, with autism spectrum disorder or language delay.
  Arms: Incredible Years Autism Spectrum and Language Delay Programme
Behavioral: First Aid for Parents — "First Aid for Parents" is a program consisting of three full day work-shops targeting communication, interaction and daily living skills for parents of children with autism spectrum disorders
  Arms: First Aid for Parents

SUMMARY:
Autism spectrum disorders (ASD) are disabling and impairing conditions affecting 1% of children in Norway. ASD is hallmarked by severe social deficit and lack of independence causing reliance on supportive systems throughout life. Parents are usually the primary caretakers and support, often throughout life. Normal parenting skills are however often ineffective due to the social dysfunction of the child with ASD. This causes high stress as the demands exceed the resources and capability of the parent. The high stress is associated to increased risk for mental health problems, divorce, unemployment and reduced quality of life. High parent stress may also reduce the effect of interventions in ASD. However, although the need is great and parental follow-up is an integral part of health care for ASD children, there is a lack of evidence for such interventions.

The current project aims to evaluate a specific parent program that is in clinical use - the Incredible Years for children with ASD - compared with a standardised treatment as usual (TAU) composed of clinical parent workshops ("first aid for parents").

The aim is to evaluate parenting interventions and promote evidence-based practice in a clinical setting. The investigators will perform a randomized controlled trial and qualitative interviews to compare the effectiveness of treatment as usual (TAU) versus a manualized parent program (IY-ASLD). The study aims to investigate if the parental program may reduce parent stress and improve parental competence and self-efficacy. Secondary goals are to investigate whether the parent program may improve quality of life for the parent and the child and have an impact on long-term child functioning and service use.

DETAILED DESCRIPTION:
Parental psychoeducation is an integral and intuitive part of health care for children with autism, but there is a lack of evidence for such interventions in general and for parental programs specifically. Studies are usually few and of poor methodological quality. Proper evaluation of parental programs is time and resource consuming. Being able to provide evidence-based parent programs is nevertheless paramount to clinical follow-up, as parents are the most crucial person in a child's life. Efficient parent programs could potentially have enormous downstream beneficial effects, as there is evidence that developmental social pragmatic treatment for parents may improve the child's functioning, but it is currently little known what kind of parent programs should be administered to whom, to what extent or in what form. Many different types of programs exist and there are some indications of what components are necessary for effect. One of the few manualized parent programs for ASD that are available in Norwegian services is the Incredible Years Autism Spectrum and Language Delay Programme (IY-ASLD©). The current project has brought together three Norwegian clinics using the IY-ASLD© to perform a multi-center RCT study. The aim is to evaluate parenting intervention in the early years for families and children with ASD.

The project hypothesizes that empowering parents to be efficient in their role as parents for children with ASD will have both short-term and long-term gains:

Short-term:

1. Improved parental stress and health
2. Improved parental competence and self-efficacy
3. Improved quality of life (QoL) for parents
4. Improved quality of life (QoL) for children

Long-term:

1. Improved child functioning
2. Reduced health service use.
3. Reduced use of alternative treatments
4. Mitigation of long-term adverse effects and disability

Main aim and primary outcome:

To evaluate the effectiveness of the IY-ASLD© vs. the TAU parenting interventions for improving primary outcome measures of lowering parental stress.

Specific hypotheses, research questions and secondary outcomes:

1. Parents in the IY-ASLD© groups will show significant improvement in a) PSI, b) paediatric quality of life and c) parent sense of competence compared with the TAU groups.
2. Children in the IY-ASLD© groups will improve more than in the TAU condition over time, with better long-term child functioning and reduced service use at 12 and 24 months.
3. To understand the subjective experiences of the parents. What are the main needs and how can and does the intervention meet these needs in the respective conditions?
4. What works for whom? Are there important moderators of effect or lack thereof? Is the child's level of functioning or level of ASD symptoms important for the effect of the intervention? Are some parental needs better met by one of the two programs?

Study design, methodology and analytic plan:

The study is planned as a multi-center RCT with a two-year follow-up. ASD is characterized by large heterogeneity and clinical complexity. Furthermore, the literature indicates there is a need for assessing and understanding the long-term effects of the intervention. These factors warrant an RCT design with long-term follow-up. As previous minor studies have all concluded that larger studies are necessary, the multi-center design is necessary to recruit the large number of families needed.

The project is planning to include minimum two PhD candidates. The first PhD project (application at NTNU pending) will focus on the baseline situation for Norwegian parents of children with ASD, using a mixed-methods approach to describe the population and validate the instruments for Norwegian use. Although the PSI, the PSOC and the PedsQL have all been used in Norway, there are no studies published on these instruments for the ASD pediatric population from Scandinavia. The qualitative interviews in the study will examine the subjective experience of the interventions, using a mixed methods approach.

The second PhD project will evaluate the effect of the intervention at T1 and T2 using the PSI as the main outcome measure (T1 and T2) as well as child outcome (PedsQL at T1 and T2, VABS at T2). Parent socio-economic status and parent competence (PSOC) as well as child function and level of ASD will be explored as mediator and moderating variables and/or covariates using structural equation modelling (SEM).

Sample size and power calculations:

Based on power calculations with statistical power of 0.8, a medium effect size (d = 0.5) and α=0.05, a sample size of minimum 64 families per condition, in total 128 families is required. Based on experience from autism follow-up in the clinic it is allowed for a drop-out rate of 20-30% and a two-parent participation rate of 80%. To allow for similar drop-out of 20-30% longitudinally and maintain power at follow up, the project aims to include 240 families. Including three sites aiming for six active condition groups over four years, the project will include an estimated number of 120 families/condition, and approximately 300-400 parental questionnaires (including PSI as the main outcome). This will allow for detection of smaller effect sizes as well as performing analyses of secondary outcomes as well as of mediating and moderating variables.

Recruitment and randomization:

During assessment of the child to determine the presence of autism, parents are interviewed at length using structured interviews. During the later feedback of the assessment to parents, the clinician at the participating sites will inform eligible parents about the project orally and in print. Information about the project will also be presented at parent organization sites, flyers and in the participating clinics. The information catalogue will also mention the project and there will be information about the project in the course catalogue at the basic parent diagnostic course.

Interested parents will be asked to register their contact details in a webtool (SurveyXact) or through direct contact/postal mail. They will be sent detailed information about the project by postal mail/e-mail (depending on their preference) and informed consent to read and sign the informed consent at their leisure.

The three participating clinics diagnose and/or treat 220-270 children with ASD every year, ensuring a large pool of families eligible for inclusion. Immigrant families are frequent in this patient group, and some of these families will thus not be eligible due to language barriers. Each clinic will run 1 or 2 IY-ASLD groups each year with the TAU condition in parallel. When 12-16 families have been recruited at a particular site, randomization to IY-ASLD© or standardized TAU will be performed.

The Incredible Years for Autism Spectrum and Language Delays program - experimental condition

The IY-ASDL program consists of 13 2 hours weekly sessions with small groups of parents of 5-7 children. The program works interactively within the parent group with video vignettes, group discussions and homework assignments between sessions to teach developmentally adapted social interaction and communication based on the child's preferences and needs.

First Aid for Parents - active control condition

The TAU condition is a three-day seminar/work-shop program, building on the content of workshops that are held at HUS as part of the regular clinical follow-up. The workshops will include communication skills, psychoeducation and approaches to daily challenges of nutrition, sleep, hygiene and daily living skills. The workshops given at HUS will be assembled and compressed to a three-day introduction program labelled "Førstehjelpen for Foreldre" (FFF; First aid for Parents). The workshops will be held once a month in the same semester as the local IY-ASDL group to ensure similar treatment periods and time from randomization and follow-up. HUS will be responsible for the development of the content and course materials for the FFF, and will also hold the program at Helse Fonna and SOH, as well as train local clinicians to hold the workshops to ensure fidelity.

User participation:

The project has involved Elisabeth Johansen from the parent organization "Autismeforeningen", from the regional "Hordaland" unit. She is a parent and as representative of the Autismeforeningen, she is in touch with many parents in different stages of their parenting.

The project is targeting user participation by design. The user feedback and evaluation of the project is essential for the delivery. Understanding the effect and experience of the parent program is part of the main outcomes of the project. Qualitative interviews with parents are part of the methodology. This part of the project is crucial to be able to go beyond the measured outcomes of the project to indicate what treatment should be offered to whom. Experiences from parents will inform future service provision to parents of children with autism.

Ethics:

The project has Regional Ethics Committee approval, nr. 188940. An important ethical challenge is the large discrepancy by the perceived need of families with children with ASD and the resources allocated to follow-up. The project aims to contribute to building better-resourced and evidenced-based care for all families living with ASD.

ELIGIBILITY:
Inclusion Criteria:

* Parent of child diagnosed with an autism spectrum disorder, age 2-6

Exclusion Criteria:

* Level of Norwegian insufficient to benefit from a parental program without the use of an interpreter
* Ongoing major crisis in the family or major disabling condition in the participating parent
* Ongoing participation in another manualized (any) parent program

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2028-10-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Parenting Stress Index - 4 Short Form | Change from Baseline Parent Stress at 6 months
  The PSI SF is a 36-item parental self-report questionnaire that assesses the stress related to interaction with the child, in relationship to the parents' personal situation and well-being. It has good psychometric properties and is one of the most commonly used questionnaires globally and is used in the corresponding studies of parental programs. To be filled in individually by all participating adults.
Parenting Stress Index - 4 Short Form | Change from Baseline Parent Stress at 18 months
  The PSI SF is a 36-item parental self-report questionnaire that assesses the stress related to interaction with the child, in relationship to the parents' personal situation and well-being. It has good psychometric properties and is one of the most commonly used questionnaires globally and is used in the corresponding studies of parental programs. To be filled in individually by all participating adults.
Parenting Stress Index - 4 Short Form | Change from Baseline Parent Stress at 30 months
  The PSI SF is a 36-item parental self-report questionnaire that assesses the stress related to interaction with the child, in relationship to the parents' personal situation and well-being. It has good psychometric properties and is one of the most commonly used questionnaires globally and is used in the corresponding studies of parental programs. To be filled in individually by all participating adults.

SECONDARY OUTCOMES:
The Vineland Adaptive Behavior Scales - Second Edition | Change from Baseline daily function of child at 18 months
  The Vineland is a measure of daily function in various domains, including social and communicative function. This measure is often used as part of the clinical assessment and level of functioning of the child, and provides standardised and age-normed scores for level of functioning in the various domains.
The Vineland Adaptive Behavior Scales - Second Edition | Change from Baseline daily function of child at 30 months
  The Vineland is a measure of daily function in various domains, including social and communicative function. This measure is often used as part of the clinical assessment and level of functioning of the child, and provides standardised and age-normed scores for level of functioning in the various domains.
The Pediatric Quality of Life Inventory (PedsQL) | Change from baseline child quality of life at 6 months
  The PedsQL is a validated questionnaire of pediatric quality of life. The parent proxy for children 2-4 years consists of 21 items in four domains: physical, emotional, social and preschool function. To be filled in individually by all participating adults.
The Pediatric Quality of Life Inventory (PedsQL) | Change from baseline child quality of life at 18 months
  The PedsQL is a validated questionnaire of pediatric quality of life. The parent proxy for children 2-4 years consists of 21 items in four domains: physical, emotional, social and preschool function. To be filled in individually by all participating adults.
The Pediatric Quality of Life Inventory (PedsQL) | Change from baseline child quality of life at 30 months
  The PedsQL is a validated questionnaire of pediatric quality of life. The parent proxy for children 2-4 years consists of 21 items in four domains: physical, emotional, social and preschool function. To be filled in individually by all participating adults.
Parenting Sense of Competence Scale (PSOC) | Change from baseline parent competence at 6 months
  The PSOC is a parent self-report questionnaire consisting of 17 items and two subscales. It has good reliability and validity and has been shown to strongly correlate with perceived parental stress in children with ASD and other developmental disorders. To be filled in individually by all participating adults.
Parenting Sense of Competence Scale (PSOC) | Change from baseline parent competence at 18 months
  The PSOC is a parent self-report questionnaire consisting of 17 items and two subscales. It has good reliability and validity and has been shown to strongly correlate with perceived parental stress in children with ASD and other developmental disorders. To be filled in individually by all participating adults.
Parenting Sense of Competence Scale (PSOC) | Change from baseline parent competence at 30 months
  The PSOC is a parent self-report questionnaire consisting of 17 items and two subscales. It has good reliability and validity and has been shown to strongly correlate with perceived parental stress in children with ASD and other developmental disorders. To be filled in individually by all participating adults.
Concomitant Treatment and Resources (Concom) | Use of services at 18 months
  The Concom is a self-report questionnaire for parents of children with ASD, to record resource and service use, including parental work reduction, alternative therapy and diet costs. To be filled in individually by all participating adults.
Concomitant Treatment and Resources (Concom) | Use of services at 30 months
  The Concom is a self-report questionnaire for parents of children with ASD, to record resource and service use, including parental work reduction, alternative therapy and diet costs. To be filled in individually by all participating adults.

CONTACTS AND LOCATIONS:
Overall Officials: Maj-Britt Posserud, MD, PhD, Principal Investigator — Haukeland University Hospital
Locations (3):
- Norway (3):
  - Haukeland University Hospital, Bergen
  - Helse Fonna, Haugesund
  - St Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No
The study includes data on a vulnerable group (non-consenting minors) and mental health, where Norwegian guidelines and rules are conservative and do not currently support sharing.

REFERENCES:
- [Background] Bearss K, Johnson C, Smith T, Lecavalier L, Swiezy N, Aman M, McAdam DB, Butter E, Stillitano C, Minshawi N, Sukhodolsky DG, Mruzek DW, Turner K, Neal T, Hallett V, Mulick JA, Green B, Handen B, Deng Y, Dziura J, Scahill L. Effect of parent training vs parent education on behavioral problems in children with autism spectrum disorder: a randomized clinical trial. JAMA. 2015 Apr 21;313(15):1524-33. doi: 10.1001/jama.2015.3150. PMID 25898050
- [Background] Bieleninik L, Posserud MB, Geretsegger M, Thompson G, Elefant C, Gold C. Tracing the temporal stability of autism spectrum diagnosis and severity as measured by the Autism Diagnostic Observation Schedule: A systematic review and meta-analysis. PLoS One. 2017 Sep 21;12(9):e0183160. doi: 10.1371/journal.pone.0183160. eCollection 2017. PMID 28934215
- [Background] Buescher AV, Cidav Z, Knapp M, Mandell DS. Costs of autism spectrum disorders in the United Kingdom and the United States. JAMA Pediatr. 2014 Aug;168(8):721-8. doi: 10.1001/jamapediatrics.2014.210. PMID 24911948
- [Background] Cappe E, Wolff M, Bobet R, Adrien JL. Quality of life: a key variable to consider in the evaluation of adjustment in parents of children with autism spectrum disorders and in the development of relevant support and assistance programmes. Qual Life Res. 2011 Oct;20(8):1279-94. doi: 10.1007/s11136-011-9861-3. Epub 2011 Feb 12. PMID 21312064
- [Background] Osborne LA, McHugh L, Saunders J, Reed P. Parenting stress reduces the effectiveness of early teaching interventions for autistic spectrum disorders. J Autism Dev Disord. 2008 Jul;38(6):1092-103. doi: 10.1007/s10803-007-0497-7. Epub 2007 Nov 20. PMID 18027079
- [Background] Reinfjell T, Diseth TH, Veenstra M, Vikan A. Measuring health-related quality of life in young adolescents: reliability and validity in the Norwegian version of the Pediatric Quality of Life Inventory 4.0 (PedsQL) generic core scales. Health Qual Life Outcomes. 2006 Sep 14;4:61. doi: 10.1186/1477-7525-4-61. PMID 16972987
- [Background] Williams ME, Hastings RP, Hutchings J. The Incredible Years Autism Spectrum and Language Delays Parent Program: A Pragmatic, Feasibility Randomized Controlled Trial. Autism Res. 2020 Jun;13(6):1011-1022. doi: 10.1002/aur.2265. Epub 2020 Jan 21. PMID 31961490
- [Background] Varni JW, Burwinkle TM, Seid M. The PedsQL as a pediatric patient-reported outcome: reliability and validity of the PedsQL Measurement Model in 25,000 children. Expert Rev Pharmacoecon Outcomes Res. 2005 Dec;5(6):705-19. doi: 10.1586/14737167.5.6.705. PMID 19807613
- [Background] Kaminski JW, Valle LA, Filene JH, Boyle CL. A meta-analytic review of components associated with parent training program effectiveness. J Abnorm Child Psychol. 2008 May;36(4):567-89. doi: 10.1007/s10802-007-9201-9. Epub 2008 Jan 19. PMID 18205039
- [Background] Lebersfeld JB, Swanson M, Clesi CD, O'Kelley SE. Systematic Review and Meta-Analysis of the Clinical Utility of the ADOS-2 and the ADI-R in Diagnosing Autism Spectrum Disorders in Children. J Autism Dev Disord. 2021 Nov;51(11):4101-4114. doi: 10.1007/s10803-020-04839-z. Epub 2021 Jan 21. PMID 33475930
- [Background] Chatham CH, Taylor KI, Charman T, Liogier D'ardhuy X, Eule E, Fedele A, Hardan AY, Loth E, Murtagh L, Del Valle Rubido M, San Jose Caceres A, Sevigny J, Sikich L, Snyder L, Tillmann JE, Ventola PE, Walton-Bowen KL, Wang PP, Willgoss T, Bolognani F. Adaptive behavior in autism: Minimal clinically important differences on the Vineland-II. Autism Res. 2018 Feb;11(2):270-283. doi: 10.1002/aur.1874. Epub 2017 Sep 21. PMID 28941213
- See also: Norwegian government document recommending parent programs for ASD follow-up — https://www.regjeringen.no/no/dokumenter/nou-2020-1/id2689221/